CLINICAL TRIAL: NCT00821314
Title: The Effect of Position (Sit/Stand up vs Supine Position) on Urge Sensation in Volunteers and in Patients With Overactive Bladder Syndrome
Brief Title: The Effect of Position on Urge Sensation in Volunteers and in Patients With Overactive Bladder Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof Dr P. E. V. van Kerrebroeck, Head of the Urology department University Hospital Maastricht, The Netherlands
Other Study IDs: MEC 08-2-128.3
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Importance of the problem OAB is a common health problem. Milsom et al. [1] randomly selected a population from six European countries. From this population, 17% of the respondents reported having OAB symptoms with 14% reporting frequency, 9% urgency, and 6% urge incontinence. The study by Milsom et al. [1] showed that OAB adversely affected the lives of the majority (65%) of the respondents who reported OAB symptoms. Chen et al. [2] also reported that the prevalence of OAB in Taiwanese women was similar to that of Western women. In the study of Chen et al.[2], the prevalence of OAB was 18.6% for the patients; perceptions and the number of OAB condition significantly increased in the elderly women (over 65 years old, 39.3%). Apart from impairing the physical health, OAB may have a tremendous effect on psychological and social well-being. Information on the symptoms and disease severity can yield important information that often complements objective measures.

Incontinence, increased urge and increased frequency of micturition affect nearly 100 million people in the western world (33 million in the US and 66 million in the European Union). These conditions are not life threatening but they seriously affect quality of life and ability to work. OAB is in some studies reported to have an incidence of up to 17 % in the western population with great consequences for the quality of life.

Economic cost The total economic cost of this group of conditions is high. In 2002 the costs in the US were approximately $12.7 billion[1] (estimated to be $17 billion and €22 billion/year in 2005). Approximately 25% of this expenditure is spent on treatment (drug therapy, clinical consultation and surgery). Of those who suffer only 28% have sought help and only half of those currently receive treatment. Less than 3% regain long lasting normal control. Therefore, these costs are an under-estimate and the problem is large.

Aetiology

DETAILED DESCRIPTION:
It is necessary to state whether correlations between objective findings and subjective perception of symptoms exist, and whether the patient's 'everyday' symptoms are reproduced during objective studies, when the results are reported. The principle aim of urodynamics is to reproduce a patient's symptoms and to provide a patho physiological explanation for them. The purposes of this study is to evaluate whether there is a relation between the position (sitting/standing up vs supine position) and the bladder sensations in both healthy volunteers and patients with OAB. Furthermore we would like to study patient perception of bladder condition and bladder filling and volumes voided as well as the functional and maximal bladder capacity in patients with OAB.

Because patients with pelvic floor dysfunction have widely varying expectations from treatment, the patient's goal for treatment is highly subjective. Therefore, strategies for assessing OAB should incorporate self-perceived disease condition.

ELIGIBILITY:
Inclusion Criteria:

* OAB must be diagnosed by their urologist using the criteria of more than 8 micturitions on three consecutive days of these three days they keep a micturation diary with a VAS score for urge sensation.
* Patients should have at least one episode of urge.

Exclusion Criteria:

* Patients with congestive heart disease and patients with a history of heart failure.
* Patients with a post voiding residual volume of more than 100 cc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of two groups. One group consist of patients with OAB. The second group consist of volunteers without micturition complaints. (25 male & 25 female)
  The second group of patients with OAB. (25 male& 25 female) Both groups will be subjected to the exact same protocol.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad S Rahnama'i', MD, Principal Investigator — University hospital Maasticht
Locations (1):
- Maastricht University Hospital, Maastricht, Limburg, Netherlands